CLINICAL TRIAL: NCT03380208
Title: Comparison of Endoscopic Visualization and CT Imaging of Head and Neck Cancers With Pathological Validation
Brief Title: Comparison of Endoscopic Visualization and CT Imaging of Head and Neck Cancers With Pathological Validation Study
Acronym: EndoscopicHN
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 17-5386
Record Dates: First submitted 2017-11-14; First posted 2017-12-21 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this clinical research is to compare new methods of identifying the locations of tumours to standard CT imaging. Analysis of the tissue removed during surgery (pathology) will be used to determine which method is more accurate. Accurately identifying the locations of tumours is especially important for radiation therapy, where the radiation needs to cover the entire tumour while minimizing the amount normal tissue that is exposed to radiation. The new method uses optical imaging (endoscopy) that can be mapped to the CT imaging using device tracking technologies. CT imaging is used to create the radiation treatment plans and so tumour locations are normally provided by CT images. The advantage of the new technology that is being tested is that it may be able to locate regions of a tumour that are at the surface of the tissue. These tumours are difficult to see using CT imaging but easy to see using optical imaging. Currently, there is no accurate way of mapping the optical imaging to the CT images used in radiation therapy.

This study will enable the investigators to test the new optical imaging by comparing the tumour that the investigators identify using CT imaging alone against using CT imaging plus the optical imaging technology. The results from this imaging will be compared to pathology findings.

DETAILED DESCRIPTION:
a CT image that includes a contrast agent that helps to identify the location of the tumour. Small markers will be placed on the participants head prior to the scan so that the investigators can align this CT image with the tracking technology used during the surgery.

The participant will be moved to the surgical table, where the surgery will proceed as it would for standard of care procedures. The tracking technology and optical imaging will be used to identify where the tumour is located at the tissue surface

* Tumour tissue and extra tissue surrounding the tumour will be removed, as would occur normally in surgery. Some markers may be placed on the tissue where it is cut. These will be helpful in matching the tissue that is removed with its location in the images.
* A second CT image will be taken immediately following the tissue removal. This will be made using an imaging device called a cone beam CT.
* In collaboration with the pathology department, whole mount tissue samples will be assessed to determine the location of tumour tissue. Using the markings on the tissue and images taken of the tissue sample after it has been removed, the location of the tumour in the tissue sample will be compared to the location of the tumour in the CT image and the location of the surface tumour determined by the optical imaging technology.
* The CT images may be analyzed by radiation oncologists, surgeons and physicists.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion in this study if they meet all of the following criteria:

Age ≥ 18 years Histologic diagnosis of oral squamous cell carcinoma Primary cancer of the H&N Intention to treat using surgery. Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Prior complete or partial radiation therapy to H&N Prior complete or partial surgery of the tumour Concurrent illness or condition that precludes subject from undergoing endoscopy or CT scanning Psychiatric or addictive disorders that preclude informed consent or adherence to protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck cancer, specifically of the oral cavity
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
CT image comparison of lesions visible in the oral cavity with pathological findings of the resected specimen. | intraop
  Relative spatial overlap of mucosal lesions in the oral cavity as detected by endoscopic imaging and gross tumor as detected by CT imaging, with confirmation of lesion pathology and location determined by whole mount pathology of the resected samples. The endoscopic imaging is co-registered to the CT image set using tracking devices embedded inside the endoscopes.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Irish, Dr., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

DOCUMENTS (1):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03380208/Prot_000.pdf